CLINICAL TRIAL: NCT05264454
Title: Effect of High-Flow Nasal Cannula on IVC Measurements Using Point of Care Ultrasound
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to Covid-19 the project will not be moving forward
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: HFNCIVC1
Record Dates: First submitted 2021-12-02; First posted 2022-03-03 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Fluid Overload
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: intervention will be blinded to those assessing the size of the IVC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0 L (Placebo Comparator): This will be the arm where the baseline IVC assessment size is conducted at
  Interventions: Device: high flow nasal cannulae
- 30 L (Active Comparator): The HFNC flow will be set at 30 L / min. The IVC size will then be assessed using a POCUS
  Interventions: Device: high flow nasal cannulae
- 60 L (Active Comparator): The HFNC flow will be set at 60 L / min. The IVC size will then be assessed using a POCUS
  Interventions: Device: high flow nasal cannulae

INTERVENTIONS:
Device: high flow nasal cannulae — The plan is to examine the effects of the size of the IVC size based upon varrying levels of high flow nasal cannulae flow
  Other Names: point of care ultrasound

SUMMARY:
The size of the inferior vena cava (IVC) using point of care ultrasound is used in resuscitation of patients who are critically ill and is now being used as a standard part of resuscitation in many clinical situations. Multiple factors can effect the size of the IVC including the type of oxygen devices the patient is currently on. In the ICU setting, the use of High Flow Nasal Cannula (HFNC) is often used to help in patients who are critically ill. There is some evidence to suggest that the use of HFNC can effect the size of the IVC measurement but the extent of the effect has not been well characterized. The purpose of this study is to determine the effect HFNC has on the size of the IVC measured using a point of care ultrasound.

DETAILED DESCRIPTION:
Shock is a state of decreased perfusion and inadequate oxygen delivery to tissues. This results in end organ damage and is associated with high morbidity and mortality, regardless of etiology. Shock associated with an infection is known as septic shock. In the intensive care unit (ICU) population, septic shock is the most common admission to the ICU and, with a mortality rate approaching 30%, is one of the leading causes of death. Early antibiotics and early intravenous fluid administration are a key component of resuscitation, but over-resuscitation with fluids is associated with adverse outcomes, including death. Therefore, methods to determine the ideal amount of fluid to administer are required.

Increasingly, the use of a bedside ultrasound, known as point of care ultrasound (PoCUS), can be used to determine the cause of shock and to help guide the ideal amount of fluid administration. One method for determining the appropriate amount of fluid to administer is the measurement of the size of the inferior vena cava (IVC). The IVC is a large vein that travels through the abdomen and delivers blood back to the heart. In a breathing patient, the size of the IVC varies with the breathing cycle. During inspiration the contraction of the diaphragm results in the generation of a negative pressure inside the chest cavity. This pressure change results in a decrease in size of the IVC during inspiration; contrary, during expiration, the IVC will be maximally distended. One of the best methods for determining fluid responsiveness using IVC is known as the IVC collapsibility index, which is defined as the [(Maximum diameter IVC-Minimum diameter) / Maximum diameter IVC] x 100. If the index is greater than 41% (range, 40%-42%), the LR ranged from 3.5 (95% CI, 1.1-15) to 9.3 (95% CI, 0.88-51) that the patient would respond to fluid.

One limitation to the use of PoCUS to assess the IVC is that the size of the vessel is affected by pressure inside the chest cavity. For example, patients who have obstructive sleep apnea (OSA) are often treated using a device called a continuous positive airway pressure (CPAP) machine. CPAP works by applying a constant amount of air pressure to prevent the soft tissues in the neck from collapsing and obstructing the airway. This constant pressure results in an increase of the chest cavity pressure which has been shown to increase the IVC diameter and a decreased IVC collapsibility index. This could result in an error in not administering fluid when the patient would benefit from it.

A patient population where this error may occur are those admitted to hospital with pneumonia. Pneumonia is the most common presentation of septic shock in critical care. Often times these patients present with septic shock as well as respiratory failure, which is treated with supplemental oxygen. Increasingly, high flow nasal cannulas (HFNC) have been used in the initial management of respiratory failure. Studies in the critically ill populations have demonstrated that, compared to conventional oxygen therapy, HFNC provides superior oxygenation and decreases the need for intubation. HFNC is a device that is able to generate very high flows (up to 60 L/min) at an adjustable FiO2 such that even at very high peak inspiratory flows (i.e. breathing in quickly), FiO2 remains consistent. These high flows generate a CPAP effect, with an approximately linear relationship of 1 cmH2O for every 10 L/min of flow. Therefore, it is possible that patients who are placed on HFNC may have an artificially enlarged IVC measurement by ultrasound.

Considering the increasing scope and utilization of PoCUS as well as HFNC in the treatment of respiratory failure, it is important to establish what effect HFNC has on POCUS IVC measurements. To date, only one study has examined the effect of HFNC on the size of IVC. This study was conducted in heart failure patients where the patients were all volume overloaded (distended IVC). The study placed patients in heart failure on HFNC on flows of 20 and 40L/min which resulted in a decrease in the IVC collapsibility index. However, no study has examined the effect of HFNC non-volume overloaded patients at 60L /min.

Our hypothesis is that the application of HFNC will increase in the size of the IVC and decrease the IVC collapsibility index in healthy patients.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* 18-40 years old

Exclusion Criteria:

* Severe lung disease (e.g. poorly controlled asthma, COPD with FEV1 <40%)
* Congestive heart failure (diastolic dysfunction, ejection fraction < 50%, severe valvular disorders)
* Renal failure
* Complete nasal obstruction or facial deformities
* BMI > 30
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Inferior vena cava maximal diameter in millimeter | 3 minutes after the intervention

SECONDARY OUTCOMES:
Inferior vena cava maximal collapsibility index | 3 minutes after the intervention
  [(Maximum diameter Inferior vena cava -Minimum diameter) / Maximum diameter Inferior vena cava] x 100

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2014 Feb 6;370(6):583. doi: 10.1056/NEJMc1314999. No abstract available. PMID 24499231
- [Background] Angus DC, van der Poll T. Severe sepsis and septic shock. N Engl J Med. 2013 Aug 29;369(9):840-51. doi: 10.1056/NEJMra1208623. No abstract available. PMID 23984731
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Background] Navaneelan T. Deaths involving sepsis in Canada. Health at a Glance. 2016;(82):11.
- [Background] Mayr FB, Yende S, Angus DC. Epidemiology of severe sepsis. Virulence. 2014 Jan 1;5(1):4-11. doi: 10.4161/viru.27372. Epub 2013 Dec 11. PMID 24335434
- [Background] Marik PE, Linde-Zwirble WT, Bittner EA, Sahatjian J, Hansell D. Fluid administration in severe sepsis and septic shock, patterns and outcomes: an analysis of a large national database. Intensive Care Med. 2017 May;43(5):625-632. doi: 10.1007/s00134-016-4675-y. Epub 2017 Jan 27. PMID 28130687
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Background] Chaves RCF, Correa TD, Neto AS, Bravim BA, Cordioli RL, Moreira FT, Timenetsky KT, de Assuncao MSC. Assessment of fluid responsiveness in spontaneously breathing patients: a systematic review of literature. Ann Intensive Care. 2018 Feb 9;8(1):21. doi: 10.1186/s13613-018-0365-y. PMID 29427013
- [Background] Perera P, Mailhot T, Riley D, Mandavia D. The RUSH exam: Rapid Ultrasound in SHock in the evaluation of the critically lll. Emerg Med Clin North Am. 2010 Feb;28(1):29-56, vii. doi: 10.1016/j.emc.2009.09.010. PMID 19945597
- [Background] Bentzer P, Griesdale DE, Boyd J, MacLean K, Sirounis D, Ayas NT. Will This Hemodynamically Unstable Patient Respond to a Bolus of Intravenous Fluids? JAMA. 2016 Sep 27;316(12):1298-309. doi: 10.1001/jama.2016.12310. PMID 27673307
- [Background] Muller L, Bobbia X, Toumi M, Louart G, Molinari N, Ragonnet B, Quintard H, Leone M, Zoric L, Lefrant JY; AzuRea group. Respiratory variations of inferior vena cava diameter to predict fluid responsiveness in spontaneously breathing patients with acute circulatory failure: need for a cautious use. Crit Care. 2012 Oct 8;16(5):R188. doi: 10.1186/cc11672. PMID 23043910
- [Background] Airapetian N, Maizel J, Alyamani O, Mahjoub Y, Lorne E, Levrard M, Ammenouche N, Seydi A, Tinturier F, Lobjoie E, Dupont H, Slama M. Does inferior vena cava respiratory variability predict fluid responsiveness in spontaneously breathing patients? Crit Care. 2015 Nov 13;19:400. doi: 10.1186/s13054-015-1100-9. PMID 26563768
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Jenkinson C, Davies RJ, Mullins R, Stradling JR. Comparison of therapeutic and subtherapeutic nasal continuous positive airway pressure for obstructive sleep apnoea: a randomised prospective parallel trial. Lancet. 1999 Jun 19;353(9170):2100-5. doi: 10.1016/S0140-6736(98)10532-9. PMID 10382693
- [Background] Au SY, Lau CL, Chen KK, Cheong AP, Tong YT, Chan LK. Hemodynamic Effects of Noninvasive Positive-Pressure Ventilation Assessed Using Transthoracic Echocardiography. J Cardiovasc Echogr. 2018 Apr-Jun;28(2):114-119. doi: 10.4103/jcecho.jcecho_53_17. PMID 29911008
- [Background] Lee CC, Mankodi D, Shaharyar S, Ravindranathan S, Danckers M, Herscovici P, Moor M, Ferrer G. High flow nasal cannula versus conventional oxygen therapy and non-invasive ventilation in adults with acute hypoxemic respiratory failure: A systematic review. Respir Med. 2016 Dec;121:100-108. doi: 10.1016/j.rmed.2016.11.004. Epub 2016 Nov 3. PMID 27888983
- [Background] Parke RL, Bloch A, McGuinness SP. Effect of Very-High-Flow Nasal Therapy on Airway Pressure and End-Expiratory Lung Impedance in Healthy Volunteers. Respir Care. 2015 Oct;60(10):1397-403. doi: 10.4187/respcare.04028. Epub 2015 Sep 1. PMID 26329355